CLINICAL TRIAL: NCT05846022
Title: Dry Needling Latent Myofascial Trigger Points and the Immediate Effect on Motor Performance: a Randomized Controlled Clinical Trial
Brief Title: Effectiveness of Dry Needling Shoulder Muscles on a Head Turning Task in Participants Aged 30-45 With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Robin Bone, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2022:098
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Neck Pain; Psychomotor Disorders
Keywords: Dry needling; Myofascial trigger points; Upper trapezius
MeSH Terms: conditions — Neck Pain; Psychomotor Disorders | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Only the physiotherapist administering the intervention of dry needling is aware of the group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): Dry needling involves the insertion of solid monofilament needles into tender points in tight muscle bands for therapeutic purposes.
  Interventions: Other: Dry Needling
- Sham needling (Sham Comparator): Shallow penetration of a solid monofilament needle into the skin alone with the "in and out" plunging movement of the needle simulated with the needle's guide tube.
  Interventions: Other: Sham Needle

INTERVENTIONS:
Other: Dry Needling — This dry needling study involves bilaterally insertion of a fine sterile needle into upper trapezius muscle fibers using a clean needling technique.
  Arms: Dry needling
Other: Sham Needle — Shallow penetration of a solid monofilament needle into the skin alone with the "in and out" plunging movement of the needle simulated with the needle's guide tube.
  Arms: Sham needling

SUMMARY:
The goal of this clinical trial is to compare the immediate effects of stimulating shoulder muscles with an acupuncture needle (dry needling) on people from thirty to forty-five years old with recurrent neck pain. The main questions this trial aims to answer are does dry needling tight shoulder muscles have an effect on:

1. the ability to turn your head with speed and accuracy,
2. your neck mobility,
3. pain,
4. the tenderness in the muscles,
5. change in your everyday function.

Participants will be asked to undergo a dry needling intervention, then participants will be asked to complete measurements before and after the including a pain scale, neck mobility, a functional questionnaire, pressure sensitivity and movement time for a repetitive head turning task. Researchers will compare the dry needling to the sham needling to see if there is a change in the measurements pre- and post-intervention.

DETAILED DESCRIPTION:
Study Design:

This is a prospective, single blind, randomized control trial with two groups. This intervention effectiveness study will utilize a pre-post clinical trial design to measure the immediate effects of the treatment of dry needling on motor performance. Specifically, dry needling bilateral upper trapezius myofascial trigger points with the primary outcome of motor performance measured by a discrete aiming head movement task called the Fitts' head turning task. Empirical evidence supports Fitts' head turning task to quantitatively measure neuromuscular functional impairments related to restricted cervical range of movement. Approval from the University of Manitoba (HS25717) ethics committee has been attained.

Purpose:

The aim of this randomized clinical trial is to measure the immediate effects of dry needling on motor function. Specifically, the effect of a single session of dry needling to shoulder/neck muscles on the performance of a repetitive head turning task.

Objectives:

1. To determine whether dry needling upper trapezius results in improved motor performance measured by the Fitts Head turning task when compared to sham needling.
2. To determine whether dry needling upper trapezius results in improved neck range of motion measured by Cervical Range of Motion instrument when compared to sham needling.
3. To determine whether dry needling upper trapezius results in a change in pain scores measured by a visual analogue scale when compared to sham needling.
4. To determine whether dry needling upper trapezius results in a change in functional ability measured by the Neck Disability Index when compared to sham needling.
5. To determine whether dry needling upper trapezius results in a reduction of pain pressure thresholds measured by pressure algometry when compared to sham needling.

Sampling:

The demographic pool will sample ages from thirty to forty-five and both genders to represent a natural clinical population. A sample size calculation was completed using G*power software based on parameters of an estimated moderate effect size of 0.75 adopted from a doctoral thesis examining the effects of cervical spinal manipulation on movement time (Gelley, 2022). A statistical power of 0.95 (equivalent to a beta = 0.05) and an alpha level of <0.05 were set. A total of thirty-six participants (18 per group) are required and will be recruited.

Participant recruitment:

Participants will be recruited from the local community of Winnipeg. Advertising will be posted in outpatient clinics, exercise gyms and studios. Outpatient practitioners (including doctors, physiotherapists, chiropractors, massage therapists) will be asked to provide the study's information to clients who meet the inclusion criteria. The practitioner involved with providing health care but not with the research will disclose the contact information to the researcher with the client's verbal consent or alternately provide the study staff's contact information. The researchers will use the personal health information/contact information for contact purposes alone. Email lists provided by clinics, gyms, studios will be sent to disseminate posters digitally. Potential participants will be sent a recruitment email with a written description of the project and the eligibility criteria. Potential participants will be asked to contact the outcome assessor via telephone or email if they are interested in participating. One reminder email will be sent to potential participants two weeks after the initial email. Another strategy will be a snowball approach, requesting potential participants to forward the invitation to any friends or colleagues that may fit the eligibility criteria. Finally, invitations to participate will be posted on social media pages as well as through researcher social media accounts (for example, Facebook, Instagram).

Data Collection Procedures:

Dry needling intervention:

Dry needling involves the insertion of solid monofilament needles into tender points in tight muscle bands for therapeutic purposes. Needles inserted into taut muscle fibres create an electrical discharge that results in twitches or muscle spasm in the targeted muscle. Dry needling is a technique that falls within the "standard of care" of physiotherapy practice, though requires training beyond basic physiotherapy education requirements. This technique may only be implemented by fully licensed physiotherapists registered on the College of Physiotherapists of Manitoba Acupuncture Roster. This intervention of dry needling involves the insertion of a fine sterile needle into upper trapezius muscle fibres bilaterally using a clean needling technique. Before the needle insertion, the muscle is pulled up and away from the thorax where it is held for the intervention. The location of the needle insertion is the taut fibres in the middle one third of the upper trapezius muscle belly. The insertion involves placing the needle's guide tube with needle tip slightly withdrawn on the patient's skin, then the index finger provides a quick tap to bypass free nerve endings below the skin, the tube is removed, then the needle is advanced into the muscle in an anterior-superior direction. The needle is plunged in the trigger point region until a local muscle twitch or sustained contraction response is achieved. An attempt to achieve four to six local muscle twitch responses will be made for therapeutic purposes. Needles and any material with body fluids are disposed of in a biohazard container.

Sham needling intervention:

There are many challenges of creating a convincing sham for an invasive technique like dry needling. The goal is to test the effectiveness of dry needling beyond the puncture's effect, thus including the puncture with the sham intervention allows the effects of needling the muscle to be isolated. Thus, the procedures for the sham needling intervention will follow the same set up as the dry needling intervention, however penetration will be shallow into the skin alone and the "in and out" plunging movement will be simulated with the needle's guide tube.

Data Collection and Analysis:

Descriptive statistical analysis will be conducted on participant demographics including gender, whether myofascial trigger points are unilateral or bilateral, age, height, weight, body mass index. The muscle's response to the needling intervention will be documented with the number of local muscle twitch response(s) observed.

Data management:

The outcome assessor will collect participant demographics and outcome measures on paper on the day of data collection, which will be stored in a locked filing cabinet within the locked laboratory space. A list of names and email addresses of participants will be kept in a secure electronic file so we can contact, send reminders to complete the survey and a summary of the results of the study. Participants' data will be collected and stored using a participant identification number. A participant contact information form will link the unique identification number to the participants' name, email address and telephone number. The participant contact information will be kept in a separate password protected computer and a password protected device. Indirect identifiers are being collected to enhance transferability of the study. Demographics of the participants will allow the research audience to consider the results with the context of the sample of the population studied. Health Insurance Portability and Accountability Act compliant software system called Jane will be used for setting up appointment dates and appointment reminders. The participant's name and email are required for this process. Data base information including the demographics, Fitts' task data, visual analogue scales, neck disability index, range of movement data, pressure algometry data and the effectiveness of blinding questionnaire will be stored initially on a password protected computer with password protected files and then will be uploaded to the College of Rehabilitation Sciences R: drive at the University of Manitoba. Consent forms and all other electronic data such as participant contact information will be uploaded to password protected files and stored on the College of Rehabilitation Sciences R: drive at University of Manitoba and will only be accessible to investigators listed in ethics submission. Once data is uploaded, the original sources will be deleted. Upon completion of the study, de-identified data will be transferred to co-investigator's R: drive for long-term storage and will be kept for five years for publication purposes.

Reporting for adverse events:

The primary investigator will report unexpected events to the academic supervisor, who will review unanticipated problems and report them to the Research Ethics board, as necessary.

While there is no guaranteed direct benefit to the participant from participation in this study, researchers are hopeful that the result of this study will support a dry needling as a clinical intervention for improving motor performance with the potential to decrease recurrent neck pain.

Change in management:

This randomized control trial is intended to meet the requirements of a master's thesis, thus there will be no change in the principal investigator. A test-retest study only requires follow-up one week post intervention, thus if recruitment goes smoothly, retaining the outcome assessor will be necessary for a short-term.

Plan for missing data:

This is a test-retest experiment that takes place within ninety minutes (about one and a half hours), so provided participants can attend the session there is not a considerable risk for missing data. Two questionnaires that will be used in the follow up to this study are The Neck Disability Index and a questionnaire to assess the success of the blinding, which will be administered by email one week after data collection and will require a nominal amount of time to complete (about five minutes). The Neck Disability Index is scored on the number of questions answered, which accommodates for missing answers. If participants neglect to answer either of the email questionnaires attempts will be made to follow up on the telephone or email. If investigators are unable to collect missing data, the questionnaires will be omitted.

Statistical analysis:

Assessment of normal distribution and assumptions of linearity, interdependence, normality, and equal variance will be undertaken for all statistical outcomes. The statistical model for the main outcome measure (the Fitts' task) will be a repeated measures analysis of variance (ANOVA). For each dependent variable analysis, the treatment group is a between subjects' factor and the other independent variables are within subject factors. The 'main effect' in terms of time, group, width, amplitude, and the interactions will be reported. Post hoc Tukey's will be employed for pairwise analysis of the interactions. Repeated measures ANOVA will be used to analyze secondary outcomes. The demographic data will undergo an independent sample t-tests for age, sex, weight, and BMI. For all statistical analysis, p values of 0.05 will be considered significant. Jamovi statistical software will be utilized to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent neck pain (with a minimum of one episode of acute neck pain corresponding to the area covered by the UT muscle in the last three months)
* a minimum of one palpable tender, taut band of muscle in the upper trapezius
* dry needling naïve
* have normal/corrected vision required for the Fitts' task
* fluent in English.

Exclusion Criteria:

* Currently experiencing an acute episode of neck pain,
* treatment to the UT or cervical spine in the last 60 days
* currently taking pain/nerve medications
* presence of upper limb neurological signs or symptoms
* any history of pathology, surgery to the cervical spine
* trauma or accident involving the cervical spine
* having general contraindications to needling (including pregnancy, acute trauma, fever or systemic infection and needle phobia)
* local contraindications at the site of the needle insertion (including local infection, open wounds, burns, inflammation, cellulitis, and undiagnosed lumps)
* precautions to needling (including history of bacterial endocarditis, heart valve replacement, pace-maker and near joint replacements).

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Fitts' Head Turning Task | 15 minutes
  The Fitts' head turning task, measures motor performance through the analysis of movement time. Fitts task experiments explore the relationship between speed and accuracy with tasks of varying degrees of difficulty- the goal of the Fitts' task is to move as quickly and accurately as possible to acquire a target. This head turning task employs a head mouse to track left and right movements with varying degrees of challenge (low, moderate, high).

SECONDARY OUTCOMES:
Pressure algometry | 5 minutes
  Pressure algometry uses an instrument to measures pressure placed on the surface of the muscle. Pain pressure thresholds are found by placing the instrument probe on the shoulder/neck muscle under investigation and applying pressure, a measurement is taken when the pressure transitions to pain.
Visual Analogue Scale (VAS) | 1 minute
  The visual analogue scale is a uni-dimensional self-report instrument used to measure the intensity of neck pain. The scale ranges from zero to ten, where zero is no pain ten is the worst pain imaginable.
Neck Disability Index (NDI) | 5 minutes
  The Neck Disability Index (NDI), a self-report questionnaire, is used to assess functional status. The test can be interpreted as a raw score with a maximum of fifty points or as a percentage. Zero points means no activity limitations and fifty points means one hundred percent complete activity limitation.
Cervical Range of Motion (CROM) | 5-10 minutes
  Range of movement is utilized as clinical measure of functional limitations for individuals with neck pain. We will use the CROM, which is the gold standard for measuring neck mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Brian MacNeil, PhD, Study Director — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No